CLINICAL TRIAL: NCT03696680
Title: Stereotactic Radiotherapy for Cerebral Metastases with Recent Hemorrhagic Signal: Phase 2 Study in 2 Steps
Brief Title: Stereotactic Radiotherapy for Cerebral Metastases with Recent Hemorrhagic Signal
Acronym: STEREO-HBM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: ANOCEF/IGCNO (Unknown); Groupement Interrégional de Recherche Clinique et d'Innovation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-A00926-49
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Hemorrhagic Brain Metastases
Keywords: hemorrhagic; brain metastases; FSRT; Stereotactic radiation therapy
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FSRT Stereotactic radiation therapy (Experimental): Each cerebral metastasis (hemorrhagic or otherwise) will be treated by radiation
  Interventions: Radiation: FSRT Stereotactic radiation therapy

INTERVENTIONS:
Radiation: FSRT Stereotactic radiation therapy — For each metastasis, dose of 30 Gy in 3 fractions at 10 Gy / fraction over 7 days

SUMMARY:
This prospective 2-stage, non-randomized Phase 2 trial evaluates the safety and efficacy of FSRT for the management of hemorrhagic brain metastases

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Performance Status 0 or 1
* Patient with less than 4 brain metastases [of a solid tumor, including melanoma, with a histologically proven diagnosis for the solid tumor; Patients who have had a metastasectomy and 1 to 3 brain metastatic lesions are eligible.
* Brain injury (s) measuring between 5 and 30 mm in diameter
* Patient eligible for stereotactic radiotherapy after a decision of the multidisciplinary committee
* Presence of intra-tumor bleeding signals on at least one brain injury before stereotactic irradiation and defined by :

  * hyperdense lesion on the non-injected CT (treatment scanner) and / or,
  * spontaneously hyperintense lesion on T1 MRI sequences without gadolinium injection and / or,
  * lesion with hypo signal on T2 sequences *
* Absence of meningeal tumor invasion
* Absence of brainstem metastasis
* DS-GPA depending on the histological type (https://brainmetgpa.com/#start):

  * Lung Adecarcinoma: DS-GPA 2 or +
  * Non-adenocarcinoma lung: DS-GPA 2.5 or +
  * Kidney: DS-GPA 2.5 or +
  * Breast: DS-GPA 2.5 or +
  * Digestive cancer: DS-GPA 3 or +
  * Melanoma: DS-GPA 1.5 or +
* Patient without concomitant anti-cancer therapy (chemotherapy, hormone therapy, anti-angiogenic or other anti-cancer treatments). Treatments should be suspended for at least 7 days before the start of FSRT radiotherapy. The treatment can be resumed 7 days after the end of radiotherapy. It's not mandatory to suspend immunotherapy
* Life expectancy estimated at over 6 months
* Patient cooperating sufficiently to perform the treatment with the use of a thermoformed mask
* Patient whose neuropsychological capacities make it possible to follow the requirements of the protocol
* Patient affiliated to a social security scheme
* Patient giving written consent

Exclusion Criteria:

* Patient with small cell lung cancer, germ cell tumors, lymphoma, leukemia and multiple myeloma
* Patient with a concomitant neurodegenerative disease
* Any symptoms not attributable to cerebral metastasis or cancerous pathology and requiring long-term use of corticosteroids (regardless of dose)
* Contraindication to brain MRI or gadolinium injection
* Hemorrhagic disorders other than intra-tumor bleeding from brain lesion (s)
* Radiosensitizing systemic disease (Neurofibromatosis ...)
* Thrombocytopenia less than 100,000 cells / mm3
* Anticoagulant treatment, and / or anti-platelet aggregation with curative et prophylaxic dose during FSRT. If treatment can be delayed for at least 5 days before starting FSRT and resumed 2 weeks after completion of FSRT, the patient is eligible.
* Hemorrhagic metastasis (s) of the brainstem
* Planning of the treatment on the target metastasis delivering a dose> 5 Gy on other metastases concomitant
* Patient with prior cerebral stereotactic irradiation
* History of total brain irradiation
* Any associated geographical, social or psychopathological condition that could compromise the patient's ability to participate in the study
* Participation in a therapeutic trial that could compromise the conduct of study
* Patient deprived of liberty or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Hemorrhagic complication rate (new hemorrhage or increase of hemorrhage) | 6 months after end of Stereotactic radiation therapy
Local tumoral response rate defined according to the recommendations of the RECIST criteria | 6 months after end of Stereotactic radiation therapy

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre de la Baie, Avranches
  - Centre François Baclesse, Caen
  - Hospices Civils de Lyon, Lyon
  - Institut de Cancérologie de Lorraine, Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lesueur P, Kao W, Leconte A, Geffrelot J, Lequesne J, Lacroix J, Brachet PE, Hrab I, Royer P, Clarisse B, Stefan D. Stereotactic radiotherapy on brain metastases with recent hemorrhagic signal: STEREO-HBM, a two-step phase 2 trial. BMC Cancer. 2020 Feb 22;20(1):147. doi: 10.1186/s12885-020-6569-1. PMID 32087691